CLINICAL TRIAL: NCT01174966
Title: Assessment of Transcutaneous Oxygen Tension and Oxygen Challenge Test in Adult Intensive Care Patients
Brief Title: Assessment of Transcutaneous Oxygen Tension/Oxygen Challenge Test in Intensive Care Unit (ICU) Patients
Acronym: ICUPtO2OCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Da wei liu, MD , Professor , Director of Department of Critical Care Medicine, Peking Union Medical College Hospital
Other Study IDs: PUMCH-ICU-LDW-OCT
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Sepsis; Shock
Keywords: oxygen challenge test; shock; mortality; Oxygen Delivery Index; cardiac output index
MeSH Terms: conditions — Sepsis; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Survivor Nonsurvivor

SUMMARY:
The lack of subcutaneous partial pressure of oxygen (PO2) rise in response to high fraction of inspired oxygen (FiO2), called the "oxygen challenge test (OCT)", was associated with higher morbidity and mortality in human subjects. Patients had negative O2 challenge test results, indicating that flow-dependent O2 consumption might have been present. Recent reports using the noninvasive transcutaneous PO2 (PtO2) and transcutaneous partial pressure of carbon dioxide probes have observed a relationship between low oxygen challenge test values to mortality and organ failure. The OCT values provides an accessible noninvasive method of detecting early shock.

To date,these studies of OCT in the ICU patients are rarely. No one has quantified OCT to CI, DO2I、ScvO2.

This study explored:

1. relationship between patient factors, hemodynamic variables, PtO2, and OCT to mortality;
2. relationship between PtO2 index, tissue oxygen index, oxygen Challenge index to CI, DO2, ScvO2.

DETAILED DESCRIPTION:
PtO2 index = PtO2/PaO2；tissue oxygen index=PtO2/FiO2；

5min OCT value = challenged 5minPtO2 - PtO2baseline；

10min OCT value= challenged 10minPtO2- PtO2baseline；

oxygen challenge index = （10minPtO2- PtO2baseline）/(10minPaO2-PaO2baseline)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Requiring a artery catheters, and pulmonary artery catheters or PiCCO-plus or central venous catheters
* FiO2<80% and SpO2>92%
* Consent informed

Exclusion Criteria:

* Not expected to live

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were sequentially admitted to the Department of Critical Care department of Peking Union Medical College Hospital from sept. of 2009 till the end of this study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 28 day after enrollmented

SECONDARY OUTCOMES:
hospital mortality | 28 day after enrollmented

CONTACTS AND LOCATIONS:
Overall Officials: dawei liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Yu M, Morita SY, Daniel SR, Chapital A, Waxman K, Severino R. Transcutaneous pressure of oxygen: a noninvasive and early detector of peripheral shock and outcome. Shock. 2006 Nov;26(5):450-6. doi: 10.1097/01.shk.0000228798.18174.6a. PMID 17047514
- [Background] Yu M, Chapital A, Ho HC, Wang J, Takanishi D Jr. A prospective randomized trial comparing oxygen delivery versus transcutaneous pressure of oxygen values as resuscitative goals. Shock. 2007 Jun;27(6):615-22. doi: 10.1097/shk.0b013e31802f0295. PMID 17505300
- [Background] Jonsson K, Jensen JA, Goodson WH 3rd, West JM, Hunt TK. Assessment of perfusion in postoperative patients using tissue oxygen measurements. Br J Surg. 1987 Apr;74(4):263-7. doi: 10.1002/bjs.1800740413. PMID 3580798
- [Background] Goeckenjan G, Strasser K. Relation of transcutaneous to arterial pO2 in hypoxaemia, normoxaemia and hyperoxaemia. Investigations in adults with normal circulation and in patients with circulatory insufficiency. Biotelemetry. 1977;4(2):77-87. PMID 610773
- [Background] Reed RL 2nd, Maier RV, Landicho D, Kenny MA, Carrico CJ. Correlation of hemodynamic variables with transcutaneous PO2 measurements in critically ill adult patients. J Trauma. 1985 Nov;25(11):1045-53. PMID 4057292